CLINICAL TRIAL: NCT01566344
Title: Reversal of Cardiomyopathy by Suppression of Frequent Premature Ventricular Complexes - A Prospective Randomized Clinical Trial
Brief Title: Reversal of Cardiomyopathy by Suppression of Frequent Premature Ventricular Complexes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL37355.068.11; METC 11-2-076 (Other: METC azm/UM)
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Heart Diseases; Cardiac Arrhythmias; Ventricular Premature Complexes; Systolic Heart Failure; Cardiomyopathies
Keywords: Premature Ventricular Complex; Cardiomyopathy; Left ventricular dysfunction; Catheter Ablation; Anti-Arrhythmic Agents; Randomized Clinical Trial
MeSH Terms: conditions — Heart Diseases; Arrhythmias, Cardiac; Ventricular Premature Complexes; Heart Failure, Systolic; Cardiomyopathies; Ventricular Dysfunction, Left

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine heart failure therapy plus PVC suppression therapy (Experimental)
  Interventions: Other: PVC suppression therapy
- Routine heart failure therapy (No Intervention)

INTERVENTIONS:
Other: PVC suppression therapy — Conventional heart failure therapy plus radiofrequency catheter ablation of PVCs as primary treatment and Amiodarone (tablets, loading dose of 600 mg per day for 4 weeks and 200 mg per day afterwards for at least 12 months) as secondary treatment in case of unsuccessful catheter ablation.
  Arms: Routine heart failure therapy plus PVC suppression therapy

SUMMARY:
Frequent monomorphic premature ventricular complexes (PVCs) may cause a cardiomyopathy (CMP) that is reversible by suppression of the ectopic focus. This study investigates whether PVC suppression therapy can improve cardiac function and clinical condition of patients with idiopathic or ischemic CMP and frequent monomorphic PVCs. For this purpose, patients will be randomized to either one of two treatment strategies: 1) conventional heart failure therapy plus PVC suppression therapy, consisting of RFCA as primary treatment and Amiodarone as secondary treatment in case of unsuccessful RFCA, or 2) conventional heart failure therapy without PVC suppression therapy.

DETAILED DESCRIPTION:
Heart failure accounts for substantial morbidity and mortality in the western world. In addition, the financial burden associated with the disease is considerable. Prognosis is generally poor and quality of life is significantly reduced. The causes of heart failure are diverse. Identification of the underlying pathophysiological mechanism is essential, because a specific patient tailored therapy may help to improve the clinical status of the individual patient. In addition, some patients may have a potentially reversible cardiomyopathy (CMP). The present study will focus on the role of frequent premature ventricular contractions (PVCs) as a cause of left ventricular (LV) dysfunction. This is a potential reversible CMP generally unknown to the cardiological society.

Frequent ventricular ectopy in patients without structural heart disease is generally thought to be a benign finding with no prognostic significance. Suppression of PVCs with anti-arrhythmic drugs or catheter ablation is therefore usually only considered when PVCs are accompanied by disabling symptoms. However, recent data suggest that frequent monomorphic PVCs (symptomatic or asymptomatic) can cause a form of CMP that may be reversible by suppression of the ectopic focus. Furthermore, the high prevalence of frequent PVCs in patients with heart disease suggests that PVC-induced CMP may be a common phenomenon. Suppression of frequent monomorphic PVCs to improve LV systolic function may therefore emerge as a new and effective treatment strategy for patients with heart failure.

Beta-blockers are safe and effective anti-arrhythmic agents and are considered the first line therapy for suppression of PVCs. Most patients with HF are already taking a beta-blocker as part of standard therapy for their underlying disease. According to international guidelines, other AADs can be used if beta-blockers are ineffective, but they have potential adverse (arrhythmic) side-effects, especially in patients with diminished LV function, and may even be contra-indicated in this patient group. In patients with LV dysfunction and frequent monomorphic PVCs that are refractory to beta-blockers, long-term drug therapy and the potential adverse (arrhythmic) side-effects of AADs can be avoided by using catheter ablation as a first alternative treatment. RFCA is already a frequently applied, widely accepted, safe, effective and potentially curative treatment for symptomatic drug refractory PVCs. It has also been safely and effectively employed in patients with tachycardia-induced CMP and patients with PVC-induced CMP. A high acute success rate of 93% and a very low PVC recurrence rate of 3% have been reported. Although recent available data suggest that elimination of the PVC source by RFCA improves LV systolic function in HF patients, it is still applied in a limited fashion for this indication because the evidence supporting this is weak. The patient series published so far were not controlled and retrospective in nature. We intend to conduct a controlled, randomized, prospective study with careful documentation and long-term follow-up to evaluate the effect of PVC suppression therapy (with RFCA as primary treatment) on cardiac systolic function in patients with CMP and beta-blocker refractory frequent monomorphic PVCs. This could establish suppression of frequent monomorphic PVCs as a potential curative treatment strategy for patients with HF.

ELIGIBILITY:
Inclusion Criteria:

1. LVEF < 50% without identifiable cause (idiopathic) or post-infarction, > 6 months.
2. Optimal conventional heart failure therapy > 3 months.
3. Frequent monomorphic PVCs on Holter monitoring.

   * Frequent = more than 15% of all QRS complexes are PVCs.
   * Monomorphic = more than 75% of PVCs have the same morphology.
4. Greater than 18 years of age.
5. Willing and capable of giving informed consent.

Exclusion Criteria:

1. Other causes of LV systolic dysfunction:

   * Significant valvular disease.
   * Untreated hypertension (blood pressure > 140 mmHg).
   * Primary CMP (HCM, ARVC, LVNC, myocarditis, stress, peripartum).
   * Secondary CMP (infiltrative, storage, toxic, neuromuscular/neurological, autoimmune).
2. Electrocardiographic PVC characteristics suggestive of a focal origin not accessible by percutaneous approach.
3. Sustained supra-ventricular arrhythmia.
4. Evidence of significant CAD (>70% stenosis of a coronary artery) on coronary angiogram (CAG) or coronary CT necessitating revascularization (PCI / CABG) in the foreseeable future.
5. Signs of current myocardial ischemia on ECG (dynamic STT segments) or during exercise testing (significant ST segment depression/elevation).
6. Myocardial infarction within the last 6 calender months prior to enrollment.
7. PCI / CABG within the last 6 calender months prior to enrollment.
8. Physical status not allowing electrophysiological study (e.g. pregnancy or severe peripheral artery disease)
9. Presence of any disease, other than the patient's cardiac disease, associated with a reduced likelihood of survival for the duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-05; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction (LVEF) | Baseline and 6 months

SECONDARY OUTCOMES:
Change in left ventricular end systolic diameter (LVESD) | Baseline and 6 months
Change in left ventricular end diastolic diameter (LVEDD) | Baseline and 6 months
Change in left ventricular end systolic volume (LVESV) | Baseline and 6 months
Change in left ventricular end diastolic volume (LVEDV) | Baseline and 6 months
Change in New York Heart Association (NYHA) functional class | Baseline and 6 months
Change in 6 minute walking distance | Baseline and 6 months
Change in quality of life (QOL) score | Baseline and 12 months
Change in serum NT-proBNP level | Baseline and 6 months
Change in premature ventricular complex (PVC) burden | Baseline and 6 months
Cost-effectiveness: costs from a health service perspective during 12 months follow-up and effectiveness measured as quality adjusted life years (QALY). | Baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Blaauw, MD, PhD, Principal Investigator — Maastricht University Medical Centre; Harry JGM Crijns, MD, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Bogun F, Crawford T, Reich S, Koelling TM, Armstrong W, Good E, Jongnarangsin K, Marine JE, Chugh A, Pelosi F, Oral H, Morady F. Radiofrequency ablation of frequent, idiopathic premature ventricular complexes: comparison with a control group without intervention. Heart Rhythm. 2007 Jul;4(7):863-7. doi: 10.1016/j.hrthm.2007.03.003. Epub 2007 Mar 12. PMID 17599667
- [Background] Takemoto M, Yoshimura H, Ohba Y, Matsumoto Y, Yamamoto U, Mohri M, Yamamoto H, Origuchi H. Radiofrequency catheter ablation of premature ventricular complexes from right ventricular outflow tract improves left ventricular dilation and clinical status in patients without structural heart disease. J Am Coll Cardiol. 2005 Apr 19;45(8):1259-65. doi: 10.1016/j.jacc.2004.12.073. PMID 15837259
- [Background] Baman TS, Lange DC, Ilg KJ, Gupta SK, Liu TY, Alguire C, Armstrong W, Good E, Chugh A, Jongnarangsin K, Pelosi F Jr, Crawford T, Ebinger M, Oral H, Morady F, Bogun F. Relationship between burden of premature ventricular complexes and left ventricular function. Heart Rhythm. 2010 Jul;7(7):865-9. doi: 10.1016/j.hrthm.2010.03.036. Epub 2010 Mar 27. PMID 20348027
- [Background] Yokokawa M, Kim HM, Good E, Chugh A, Pelosi F Jr, Alguire C, Armstrong W, Crawford T, Jongnarangsin K, Oral H, Morady F, Bogun F. Relation of symptoms and symptom duration to premature ventricular complex-induced cardiomyopathy. Heart Rhythm. 2012 Jan;9(1):92-5. doi: 10.1016/j.hrthm.2011.08.015. Epub 2011 Aug 17. PMID 21855522
- [Background] Sarrazin JF, Labounty T, Kuhne M, Crawford T, Armstrong WF, Desjardins B, Good E, Jongnarangsin K, Chugh A, Oral H, Pelosi F, Morady F, Bogun F. Impact of radiofrequency ablation of frequent post-infarction premature ventricular complexes on left ventricular ejection fraction. Heart Rhythm. 2009 Nov;6(11):1543-9. doi: 10.1016/j.hrthm.2009.08.004. Epub 2009 Aug 5. PMID 19879531
- [Background] Blaauw Y, Pison L, van Opstal JM, Dennert RM, Heesen WF, Crijns HJ. Reversal of ventricular premature beat induced cardiomyopathy by radiofrequency catheter ablation. Neth Heart J. 2010 Oct;18(10):493-8. doi: 10.1007/BF03091821. PMID 20978594
- [Background] Niwano S, Wakisaka Y, Niwano H, Fukaya H, Kurokawa S, Kiryu M, Hatakeyama Y, Izumi T. Prognostic significance of frequent premature ventricular contractions originating from the ventricular outflow tract in patients with normal left ventricular function. Heart. 2009 Aug;95(15):1230-7. doi: 10.1136/hrt.2008.159558. Epub 2009 May 7. PMID 19429571
- [Background] Kanei Y, Friedman M, Ogawa N, Hanon S, Lam P, Schweitzer P. Frequent premature ventricular complexes originating from the right ventricular outflow tract are associated with left ventricular dysfunction. Ann Noninvasive Electrocardiol. 2008 Jan;13(1):81-5. doi: 10.1111/j.1542-474X.2007.00204.x. PMID 18234010
- [Background] Duffee DF, Shen WK, Smith HC. Suppression of frequent premature ventricular contractions and improvement of left ventricular function in patients with presumed idiopathic dilated cardiomyopathy. Mayo Clin Proc. 1998 May;73(5):430-3. doi: 10.1016/S0025-6196(11)63724-5. PMID 9581582
- [Background] Yarlagadda RK, Iwai S, Stein KM, Markowitz SM, Shah BK, Cheung JW, Tan V, Lerman BB, Mittal S. Reversal of cardiomyopathy in patients with repetitive monomorphic ventricular ectopy originating from the right ventricular outflow tract. Circulation. 2005 Aug 23;112(8):1092-7. doi: 10.1161/CIRCULATIONAHA.105.546432. Epub 2005 Aug 15. PMID 16103234
- [Background] Taieb JM, Maury P, Shah D, Duparc A, Galinier M, Delay M, Morice R, Alfares A, Barnay C. Reversal of dilated cardiomyopathy by the elimination of frequent left or right premature ventricular contractions. J Interv Card Electrophysiol. 2007 Nov;20(1-2):9-13. doi: 10.1007/s10840-007-9157-2. Epub 2007 Oct 17. PMID 17940858
- [Background] Kennedy HL, Whitlock JA, Sprague MK, Kennedy LJ, Buckingham TA, Goldberg RJ. Long-term follow-up of asymptomatic healthy subjects with frequent and complex ventricular ectopy. N Engl J Med. 1985 Jan 24;312(4):193-7. doi: 10.1056/NEJM198501243120401. PMID 2578212